CLINICAL TRIAL: NCT04261764
Title: Fasting-mimicking Diet Combined With Traditional Chinese Medicine for Phlegm-dampness Type Obesity Patients(FASTAR): a Randomized Controlled Study
Brief Title: Fasting-mimicking Diet Combined With Traditional Chinese Medicine for Phlegm-dampness Type Obesity Patients
Acronym: FASTAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yuanqi Zhao,MD, Principal Investigator, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCM-FMD
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Obesity
Keywords: Obesity; Fasting-mimicking diet; Chinese medicine
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM-FMD (Experimental): Fasting-Mimicking Diet Combined With a "Dispelling Dampness" Meal Replacement Apply fastening-mimicking diet combined with a "dispelling dampness" meal replacement. For the convenience of implementation, a cycle of 4 weeks. The first 5 days of each cycle is the calorie restriction stage (daily calorie about 800kcal). The traditional Chinese medicine with dampness effect is used as the main source of calories in this stage. The normal diet is carried out under the guidance of a professional dietitian for the next 23 days. Study for 12 weeks.
  Interventions: Device: Fastening-mimicking diet combined with a "dispelling dampness" meal replacement
- Normal diet (Placebo Comparator): Carrying out normal diet under the guidance of a dietitian, for 12 weeks.
  Interventions: Other: Normal diet

INTERVENTIONS:
Device: Fastening-mimicking diet combined with a "dispelling dampness" meal replacement — Apply fastening-mimicking diet combined with a "dispelling dampness" meal replacement. For the convenience of implementation, a cycle of 4 weeks. The first 5 days of each cycle is the calorie restriction stage (daily calorie about 800kcal). The traditional Chinese medicine with dampness effect is used as the main source of calories in this stage. The normal diet is carried out under the guidance of a professional dietitian for the next 23 days. Study for 12 weeks.
  Arms: TCM-FMD
Other: Normal diet — Carrying out normal diet under the guidance of a dietitian.
  Arms: Normal diet

SUMMARY:
The primary aim of this study is to is to determine if a diet (TCM-FMD) which combine fasting-mimicking diet (FMD) with "dispelling dampness" meal replacement (a meal replacement made up of traditional Chinese medicine) is the effective dietary strategy for treatment of phlegm-dampness type overweight/obese patients. A three months randomized trial will be used to observe weight loss generated by TCM-FMD. And a group keeping a normal diet will be set as a blank control. Through comparison, we aim at examining the effects of interventions on weight and the diversity and abundance of intestinal flora .

DETAILED DESCRIPTION:
Background: Fasting-mimicking Diet (FMD) is a plant-based diet designed to attain fasting-like effect, firstly proposed on 2015. It requires people to limit calorie intake for 5 continuous days, and then return to their normal diet after completion about 25 days until the next cycle. In a clinical trial, three FMD cycles reduced body weight, trunk and body fat, and reduced blood pressure, fasting blood glucose, triglycerides and total cholesterol. On the other hand, in the theory of physique of TCM theory, overweight/obesity is usually considered to be phlegm-dampness type.

Objective: We assume that using medicinal-edible plants which was considered to dispel dampness(such as fuling, shanyao, etc.) as FMD's proprietary formulations can enhance the effect of FMD on improve people's characteristic features of metabolic syndrome.

Methods: A 12-week, single-center, pilot study will be conducted to test the study objectives. A new diet is carried. It is a fasting-mimicking diet combined with a "dispelling dampness" meal replacement. Because the theory of applying traditional Chinese medicine combined with FMD, which one the main ingredient of the "dispelling dampness" meal package is Chinese Herbal Medicine such as shaoyao, yiyiren, and chixiaodou, etc. At the same time, a group of normal diets was also designed as a blank control group.

Outcomes: The primary outcome measure for the study was changes in the diversity and abundance of intestinal flora, the number of Firmicutes, Bacteroides and the ratio of Firmicutes/Bacteroides; secondary outcome measures included: weight, BMI, waist circumference, blood pressure, triglycerides, total cholesterol and fasting blood glucose, etc. Both groups were subjected to caloric restriction (5 days, daily calorie about 800kcal) and normal diet (dietitian for healthy diet guidance), and the blank control group was given a normal diet.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as overweight / obesity according to the "China Adult Obesity Prevention and Treatment Expert Consensus"
* Diagnosis as phlegm-dampness type according to the "Traditional Chinese Medicine Classification and Judgment" scale published by the Chinese Medicine Association
* 18 years old ≤ age ≤ 65 years old
* Signed the informed consent

Exclusion Criteria:

* Those who have special food requirements or having a history of food allergies
* Those who have history of previous diabetes, or body weight loss, BMI ≤ 18
* Those who have had cardiovascular and cerebrovascular events within half a year, or who have a major history of surgery
* Pregnant or lactating woman
* Those who have severe primary diseases such as liver or kidney diseases, as well as abnormalities in the hematopoietic system and mental disorders
* Those who need to take special drugs (such as hormones)
* Those who refuse to provide information required for research (such as personal information, blood samples, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-11-12 (Estimated); Study Completion 2022-02-12 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota Gut microbiota | Change from baseline to week 12
  Changes in the diversity and abundance of intestinal flora, the number of Firmicutes, Bacteroides and the ratio of Firmicutes/Bacteroides

SECONDARY OUTCOMES:
Body morphology indicators | Change from baseline to week 12
  Changes in body morphology indicators (weight, BMI, waist circumference, body fat percentage, skeletal muscle weight, etc.)
Fasting glucose | Change from baseline to week 12
  Changes in fasting blood glucose
Blood pressure | Change from baseline to week 12
  Changes in blood pressure
Blood lipids | Change from baseline to week 12
  Changes in blood lipids

CONTACTS AND LOCATIONS:
Locations (1):
- Yuanqi physical Zhao, Guangzhou, Guangdong, China